CLINICAL TRIAL: NCT04666545
Title: Multidisciplinary Support To Access Living Donor Kidney Transplant (MuST AKT)- A Pilot Randomized Controlled Trial
Brief Title: Multidisciplinary Support To Access Living Donor Kidney Transplant-Pilot
Acronym: MuST AKT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: University Hospital Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pro00097902
Record Dates: First submitted 2020-11-23; First posted 2020-12-14 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Living Donor Kidney Transplantation

STUDY DESIGN:
Intervention Model Description: Pilot parallel block randomized controlled trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This arm will receive the MuST AKT intervention, which is a multidisciplinary, tailored person-centered behavioural intervention designed to "help and enable" the potential kidney transplant recipients to achieve what is required to receive a living donor kidney transplantation.
  Interventions: Behavioral: MuST AKT
- Usual Care (control) (No Intervention): In the usual care (control) condition, participants will go through the current standard of care, which is a social worker assessment.

INTERVENTIONS:
Behavioral: MuST AKT — A behavioural intervention designed to help participants identify and communicate with their social network about living kidney donation.
  Arms: Intervention

SUMMARY:
For patients with kidney failure the two treatment options are kidney transplantation or dialysis. Transplantation offers longer survival, better quality of life and provides cost savings for the health system (>$60,000/year per patient). Unfortunately, there are not enough organs available and 20% of patients die on dialysis waiting for a deceased donor kidney.

Living kidney donation is a safe and proven treatment that leads to even better patient and health system outcomes than deceased donor kidney transplant. The Kidney Health Strategic Clinical Network (KH-SCN) identified increasing living kidney donation as a priority and in 2015 established the Living Donor Kidney Transplant Working Group (LDKTWG) comprised of patients, donors, health care professionals, researchers, and administrators. In an evidenced review published by the investigators, the intervention with the best evidence and greatest impact was personalized support provided by a multidisciplinary team to inform and educate the patients' social network. This intervention increased living kidney donations by 34%. The investigators confirmed through a province wide survey that many patients with kidney failure are unable to find a living kidney donor and find it difficult to approach potential donors due to lack of skills, supports, and resources and these issues are particularly apparent in vulnerable populations. The investigators have developed the Multidisciplinary Support To Access living donor Kidney Transplant (MuST AKT) intervention to support patients in identifying and communicating with their social networks. The investigators will test the effectiveness of this intervention.

DETAILED DESCRIPTION:
Living donor kidney transplantation is the optimal treatment for end-stage kidney disease patients, dramatically improving survival and quality of life, providing significant cost saving compared with dialysis, reducing the demand for deceased donor transplants and the pressure to increase dialysis capacity and infrastructure. Outcome data shows that only 16% of Canadians on dialysis survive past 10 years, whereas up to 74% of Canadians with a kidney transplant have a functioning kidney after 10 years. The ideal treatment trajectory is to avoid dialysis entirely and receive a living donor transplant prior to dialysis (pre-emptive), which unfortunately only occurs in 10.5% of eligible patients.

Patients with end-stage kidney disease report being overwhelmed with other issues (loss of work, family stress, fear of dialysis) and lack the skills needed to comfortably engage potential living donors - many feel uncomfortable doing so and do not know how to start. The purpose of this research is to test an intervention designed to support patients identification of potential donors and communication with their social network and ultimately increase the number of living donor kidney transplantations.

Justification:

The rate of living kidney donor transplantation is lower in Alberta compared to other provinces in Canada. As the rate of kidney failure has increased over the past few years in Alberta, it is necessary to improve and facilitate the process of living kidney donor transplantation for better patient care.

Primary Objective:

The primary objective of this study is to examine the efficacy of the MuST AKT program to facilitate patients' identification of potential living kidney donors compared to usual care.

Hypothesis:

The investigators hypothesize that the MuST AKT program will increase the proportion of participants with at least one potential living kidney donors who started evaluation (intervention vs control).

Additional Objectives:

The secondary objective is to evaluate patient outcome improvement by collecting Patient Reported Outcome Measures (PROMs) to assess the proportion of patients who find at least one potential living donor.

The tertiary objective is to evaluate patient experience by collecting Patient Reported Experience Measures (PREMs) to determine whether participants recommend this program to other patients and to what extent this program gave them confidence for finding a potential living kidney donor.

The quaternary objective is to evaluate the feasibility of this program by assessing consent rate, attendance, adherence, and drop-out.

Research Methods/Procedures:

This is a pilot parallel randomized controlled trial with a qualitative interview component. The intervention condition will receive a multidisciplinary, tailored person-centered intervention over three months (MuST AKT program), and the control condition will receive the current standard of care (social worker assessment).

Patients who have been referred for kidney transplantation assessment in Edmonton will be contacted during a standard care kidney transplant education session or over the telephone if patients have completed the transplant education and are on the deceased kidney donor wait-list. Patients who expressed interest will be contacted via telephone by a member of the research team to seek their consent, complete the initial screening assessment to confirm their eligibility and enrolment, and then complete a baseline questionnaire. Then participants will be randomized to either the intervention or control condition, using predetermined randomly-generated (by Stata MP 15·1) permuted blocks of 4 and 6. Assignment to condition will be concealed by the database up until the point of assignment. Participants in the intervention condition will receive the MuST AKT program and participants in the control condition will receive usual care. Consent rate, attendance, adherence, and drop-out will be tracked during enrollment and the duration of the intervention. Upon completion of the intervention (or usual care), participants will complete a post-intervention questionnaire to assess PREMs. Participants in the intervention condition will be contacted after they have completed the post-questionnaire to participate in a qualitative interview lasting approximately 40 minutes. Kidney transplant status will be tracked for a period of 24 months post-intervention. Participants in the intervention condition who do not have a potential donor come forward after 12 months will be contacted to complete an additional interview to explore factors contributing to their lack of success, which will last approximately 40 minutes.

Intervention Condition: MuST AKT is a multidisciplinary, tailored person-centered intervention aimed to support participants identification of potential donors and communication with their social network. A one-on-one introductory session will be followed by three 'one-on-one' sessions (A, B and C) and a final session D with participants family and friends (potential donors and advocates) identified in session A. All group and individual sessions will be arranged virtually during the COVID-19 pandemic, and may be held either virtually or in-person, at the participants discretion, in the event that the COVID-19 pandemic concludes and physical distancing requirements have been eliminated. Each education session will take approximately 90 minutes. Sessions will be facilitated by a trained licensed social worker, coordinator or social media expert with extra training in kidney disease, transplantation, living kidney donation, counselling and interviewing, and patient confidentiality.

Usual care (control condition): In the control condition, participants will go through the current standard of care, which is a social worker assessment. If the intervention is successful in the definitive RCT (to be conducted later) and approved by Alberta Health Services as the 'new standard of care', people in control condition will be contacted and given the option to participate in the MuST AKT program.

Additional interviews with separate informed consent procedures:

(Patients) If, during recruitment for the study, the individual indicates they do not want to participate, or if participants drop-out of the study, a research team member will invite them participate in a 20-40 minute interview to understand barriers to participation in the study.

(Friends and family of patients) Friends and family members of participants who take part in session D will be invited to participate in an interview approximately 40 minutes long which aims to explore their experiences of group session D.

Plan for Data Analysis - Quantitative:

All analyses will be completed in Stata/MP 17.0 (www.stata.com), using an intention-to-treat approach. The investigators will use the Fisher's exact tests (dichotomous outcomes) and t-tests or Wilcoxon rank-sum tests (continuous outcomes data), as appropriate.

Our primary analyses (of our primary and secondary outcomes #1-4) will pool data from both the current and the definitive trials. In secondary analyses, the investigators will generate within trial results to investigate potential heterogeneity of intervention delivery.

Plan for Data Analysis - Qualitative Telephone interviews will be conducted using semi-structured interview guides. Data will be analyzed using a thematic analysis approach, whereby common themes that emerge from the data are documented. The qualitative software NVivo-12 will be used in the analysis.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* No obvious contraindication to kidney transplantation
* Completed 'introduction to kidney transplant' module

Exclusion Criteria:

* Potential Living Kidney Donor identified
* Previously received organ transplant
* Candidate for multi-organ transplant
* Stanford Integrated Psychosocial Assessment for Transplant (SIPAT) Score > 20
* Rapid Estimate of Adult Literacy in Medicine (REALM-66) score < 19 (illiterate in English)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Living Kidney Donor Evaluation Started | 12 months
  Proportion of participants with at least one potential donor who started evaluation

SECONDARY OUTCOMES:
Living Kidney Donor Transplantation | 24 months
  Proportion of living kidney donor transplantations
Contact Living Donor Services | 12 months
  Proportion of participants with at least one potential donor who contacted living donor services
Living Kidney Donor Evaluation Completed | 12 months
  Proportion of participants with at least one potential donor who completed evaluation
Identified potential advocates | From date of first to last documented session, an average of 3 months
  Number of participants who found at least one potential advocate

OTHER OUTCOMES:
Participant recommendation | At date of last documented session, an average of 3 months
  Proportion of patients who recommend the program they receive
Perception of program effectiveness (1 item developed for this study) | At date of last documented session, an average of 3 months
  Participants rate the following prompt on a scale from 1(completely disagree) to 7 (completely agree): "This program was effective at finding me a living kidney donor". A higher score indicates a better outcome.
Self-efficacy for approaching a potential donor as assessed by 1 item developed for this study: "How confident are you that you can talk to a friend or family member about being a potential living kidney donor?" | 3 months (length of intervention)
  Participants rate the following prompt on a scale from 0 (not at all confident) to 100 (complete confidence): "How confident are you that you can talk to a friend or family member about being a potential living kidney donor?". Higher scores indicate a better outcome.
Self-efficacy for finding a living kidney donor assessed by 1 item developed for this study: "How confident are you that you can find a potential living kidney donor?" | 3 months (length of intervention)
  Participants rate the following prompt on a scale from 0 (not at all confident) to 100 (complete confidence): "How confident are you that you can find a potential living kidney donor?". Higher scores indicate a better outcome.
Consent rate | From start date to end date of study recruitment, up to 1 year
  proportion of eligible participants who consented
Drop-out rate (overall study) | From date of enrollment to date of last documented session, an average of 4 months
  proportion of participants who withdrew consent
Intervention session completion | From date of first to last documented session, an average of 3 months
  proportion of participants who completed each session in the intervention
Intervention session drop-out | From date of first to last documented session, an average of 3 months
  proportion of intervention sessions postponed or not completed
Identified donor and advocate | From date of first to last documented session, an average of 3 months
  proportion of participants who identify at least one donor and/or advocate
Conversation started | From date of first to last documented session, an average of 3 months
  proportion of participants who started a conversation with at least one potential donor
Advocate and donor attendance at last intervention session | At date of last documented session, an average of 3 months
  total number of people who attend the last intervention session

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Shojai, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Selzler AM, Davoodi PM, Klarenbach S, Lam NN, Smith T, Ackroyd A, Wiebe N, Corradetti B, Ferdinand S, Iyekekpolor D, Smith G, Verdin N, Bello AK, Wen K, Shojai S; Multidisciplinary Support To Access living donor Kidney Transplant (MuST AKT) Research Group. Multidisciplinary Support To Access living donor Kidney Transplant (MuST AKT): A Clinical Research Protocol for a Pilot Randomized Controlled Trial to Increase Living Kidney Donation. Can J Kidney Health Dis. 2023 Oct 30;10:20543581231205340. doi: 10.1177/20543581231205340. eCollection 2023. PMID 37920779